CLINICAL TRIAL: NCT04742049
Title: The Effects of Telerehabilitation on Peripheral Muscle Function, Physical Activity Level and Sleep Quality in Pediatric Cystic Fibrosis Patients Having Social Isolation Due to Pandemic
Brief Title: The Effects of Telerehabilitation on Muscle Function, Physical Activity and Sleep in Cystic Fibrosis During Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Kılıç, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-20058
Record Dates: First submitted 2021-01-17; First posted 2021-02-05 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis; Covid19; Social Isolation
Keywords: exercise; sleep; cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis; COVID-19; Social Isolation; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Telerehabilitation based exercise training will be given to the study group.
  Interventions: Other: Telerehabilitation-based
- Exercise brochure (Experimental): Exercise training will be provided by sending a document to the control group
  Interventions: Other: Follow-up based

INTERVENTIONS:
Other: Telerehabilitation-based — 15 pediatric cystic fibrosis patients who are at home during the self- isolation process due to the COVID-19 pandemic will be included in this group. Online exercise training protocol will be apply for patients. Each training protocol was planned as 30 minutes for 3 days a week for 6 weeks with a physiotherapist. Exercise protocol will start with the warm-up exercises and finish with cooling exercises.
  Arms: Telerehabilitation
Other: Follow-up based — 15 pediatric cystic fibrosis patients who are at home during the self- isolation process due to the COVID-19 pandemic will be included in this group. An exercise document including the same exercise protocol in study group will be sent the patients. Patients will be called by the physiotherapist once a week for follow-up. .
  Arms: Exercise brochure

SUMMARY:
The aim of this study is to evaluate the peripheral muscle function, sleep disorders and physical activity level in children with cystic fibrosis who are physically inactive at home due to social isolation and to examine the effect of the 6-week online exercise protocol.

DETAILED DESCRIPTION:
Considering the new coronavirus (COVID-19) pandemic global information, some patient populations have been identified at higher risk of this pandemic like older age, hypertension, cardiovascular and respiratory diseases. Self- isolation is recommended for preventive strategy in cystic fibrosis patients. Long-term social isolation and school closure can have negative effects on childrens' physical and mental health. Due to social isolation childrens are less physical active, have longer screen exposure and irregular sleep patterns.

There is no study to evaluate the the peripheral muscle function, sleep disorders and physical activity level and examine the effects of exercise training in children with cystic fibrosis in social isolation due the COVID-19 pandemic.

This study will be included children with cystic fibrosis who had stabile conditions Patients' peripheral muscle function, sleep quality and physical activity level will be assess and record at beginning, after the twelve and eighteen session.

ELIGIBILITY:
Inclusion Criteria:

* People who diagnosed cystic fibrosis disease at stabile conditions.
* Volunteering to participate in the study,
* Having a social isolation due to COVID-19 pandemic
* Having forced expiratory volume at one second (FEV1) %> 40 % at last pulmonary function test.

Exclusion Criteria:

* Being diagnosed with acute pulmonary exacerbation at the time of study and / or within the last month.
* having a diagnosed with COVID-19 before or during the study
* Being physically or perceptually competent to exercise
* Patients with allergic bronchopulmonary aspergillosis (ABPA) who were treated with systemic steroid therapy
* Patients who were not complete the exercise training ability.
* Having FEV1 %< 40% at pulmonary function test.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
1 minute sit to stand test (STS) repetitions | before exercise training
  number of sit to stand for one minute is recorded
1 minute sit to stand test (STS) repetitions | one month
  number of sit to stand for one minute is recorded
1 minute sit to stand test (STS) repetitions | six week
  number of sit to stand for one minute is recorded

SECONDARY OUTCOMES:
sleep quality assessment | before exercise training
  Sleep quality will be evaluated by Epworth Sleepiness Scale and Pediatric Sleep Questionnaire (PSQ). Epworth Sleepiness Scale evaluates persons' daytime sleepiness and scores ranged from 0-24. Higher scores indicate higher daytime sleepiness. PSQ consist of 22 items that evaluate the frequency and severity of snoring during sleep, apnea at night during sleep hyperactivity and other pediatric obstructive sleep apnea symptoms. Responses to the items are as "yes", "no" and "I don't know" which are scored as 1, 0 and missing respectively. Total score of PSQ is the mean of the scores of all items excluding the missing items.
sleep quality assessment | six week
  Sleep quality will be evaluated by Epworth Sleepiness Scale and Pediatric Sleep Questionnaire (PSQ). Epworth Sleepiness Scale evaluates persons' daytime sleepiness and scores ranged from 0-24. Higher scores indicate higher daytime sleepiness. PSQ consist of 22 items that evaluate the frequency and severity of snoring during sleep, apnea at night during sleep hyperactivity and other pediatric obstructive sleep apnea symptoms. Responses to the items are as "yes", "no" and "I don't know" which are scored as 1, 0 and missing respectively. Total score of PSQ is the mean of the scores of all items excluding the missing items.
physical activity level | before exercise training
  Physical activity level will be evaluated by Physical Activity Questionnaire. Physical Activity Questionnaire is composed ten questions that evaluate the physical activity status for the last seven days. Each question, except last question is evaluated on a 5-point scale and there is an activity score between 1-5. "1" indicates low physical activity, "5" indicates high physical activity.
physical activity level | six week
  Physical activity level will be evaluated by Physical Activity Questionnaire. Physical Activity Questionnaire is composed ten questions that evaluate the physical activity status for the last seven days. Each question, except last question is evaluated on a 5-point scale and there is an activity score between 1-5. "1" indicates low physical activity, "5" indicates high physical activity.
crunch repetitions | before exercise training
  number of crunch completed is recorded
crunch repetitions | one month
  number of crunch completed is recorded
crunch repetitions | six week
  number of crunch completed is recorded
squat repetitions | before exercise training
  number of squats completed is recorded
squat repetitions | one month
  number of squats completed is recorded
squat repetitions | six week
  number of squats completed is recorded
push-up repetitions | before exercise training
  number of push-ups completed is recorded
push-up repetitions | one month
  number of push-ups completed is recorded
push-up repetitions | six week
  number of push-ups completed is recorded
plank duration | before exercise training
  duration of keeping plank position is recorded
plank duration | one month
  duration of keeping plank position is recorded
plank duration | six week
  duration of keeping plank position is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Dogru-Ersoz, Professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No